CLINICAL TRIAL: NCT02646722
Title: Relation Between Withdrawal Movement on Rocuronium Injection and Emergence Agitation and Pain in Preschool Ages: Observational Study
Brief Title: Relation Between Withdrawal Movement for Rocuronium and Emergence Agitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Go Un Roh, principal investigator, Ajou University School of Medicine
Other Study IDs: AJIRB-MED-OBS-15-169
Record Dates: First submitted 2015-12-28; First posted 2016-01-06 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No pain: patients show no pain on rocuronium injection
- mild pain: patients move a hand only on rocuronium injection
- moderate pain: patients move a arm on rocuronium injection
- severe pain: patients show generalized movement because of pain

SUMMARY:
Rocuronium results in burning pain on injection site. It can be reduced by local anesthetics or opioid, but still some patients, especially in children, show withdrawal movement for pain. This might resulted from individual pain sensitivity.

Emergence agitation (EA) in children is quite frequent postoperatively and is known to be associated with postoperative pain. If a patient is susceptible to postoperative pain, he or she would have high probability of EA postoperatively. Therefore, the investigators explore the relation of withdrawal movement of rocuronium and EA.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I, II

Exclusion Criteria:

* Intravenous cannulation other than a hand or an upper arm with 24 gauge catheter

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients scheduled for inguinal hernioplasty in university hospital
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
emergence agitation (Watcha scale) | 1 min after postanesthesia care unit (PACU) admission
  Watcha scale

SECONDARY OUTCOMES:
Pain (FLACC scale) | 1. 1 min after postanesthesia care unit (PACU) admission 2. 10 min after PACU admission 3. 20 min after PACU admission 4. 30 min after PACU admission 5. 40 min after PACU admission
  FLACC scale (Face, Leg, Activity, Cry, Consolability)
emergence agitation (Watcha scale) | 2. 10 min after PACU admission 3. 20 min after PACU admission 4. 30 min after PACU admission 5. 40 min after PACU admission

CONTACTS AND LOCATIONS:
Overall Officials: Go Un Roh, MD, Principal Investigator — Ajou University School of Medicine

IPD SHARING:
Plan to Share IPD: No